CLINICAL TRIAL: NCT06799494
Title: Comparing the Antibody and B Cell Responses Induced by 1- or 2-dose 9-valent HPV (9vHPV) Vaccination in Healthy Adults
Brief Title: HPV Vaccine Reduced Dose
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Erin Scherer, PhD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00008623
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: HPV
Keywords: HPV Prevention; HPV Vaccine; Immune responses
MeSH Terms: interventions — Papillomavirus Vaccines; Lidocaine; Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- One dose of the 9-valent HPV vaccine (Experimental): Participants will receive one dose of the 9-valent HPV (9vHPV) vaccine by intramuscular injection on Day 0.
  Participants will be asked to donate blood samples for immunologic testing at screening (from Day -60 to -1), on Day 0 (before vaccination), 7±1, 30±5, 180±5 (before vaccination; Visit 5), Visit 5 + 7±1 days, Visit 5 + 30±5 days, 365±14, 730±14, 1095±14, 1460±14, 1825±30 (Visit 15), and ≥84 days from Visit 15 (Optional Visit 17).
  Axillary lymph node sampling by fine needle aspiration (FNA) will be done 3 times per group on Day 30±5, 180±5 (Visit 5), Visit 5 + 30±5 days.
  Bone marrow sampling will be done for all groups at Days 730±14 and 1825±30.
  Interventions: Biological: Gardasil-9; Drug: Lidocaine injection; Drug: Lorazepam
- Two doses of the 9-valent HPV vaccine (Active Comparator): Participants will receive two doses of the 9vHPV vaccine on Day 0 and a second dose 6 months later.
  Participants will be asked to donate blood samples for immunologic testing at screening (from Day -60 to -1), on Day 0 (before vaccination), 7±1, 30±5, 180±5 (before vaccination; Visit 5), Visit 5 + 7±1 days, Visit 5 + 30±5 days, 365±14, 730±14, 1095±14, 1460±14, 1825±30 (Visit 15), and ≥84 days from Visit 15 (Optional Visit 17).
  Axillary lymph node sampling by fine needle aspiration (FNA) will be done 3 times per group on Day 30±5, 180±5 (Visit 5), Visit 5 + 30±5 days.
  Bone marrow sampling will be done for all groups at Days 730±14 and 1825±30.
  Interventions: Biological: Gardasil-9; Drug: Lidocaine injection; Drug: Lorazepam

INTERVENTIONS:
Biological: Gardasil-9 — The 9-valent HPV VLP vaccine is a sterile liquid suspension prepared by combining the adsorbed VLPs of each HPV type and additional amounts of the aluminum-containing adjuvant and the final purification buffer. The 9-valent HPV vaccine, or Gardasil-9, is a sterile suspension for intramuscular administration. Each 0.5-mL dose of the vaccine also contains approximately 500 mcg of aluminum (provided as AAHS), 9.56 mg of sodium chloride, 0.78 mg of L-histidine, 50 mcg of polysorbate 80, 35 mcg of sodium borate, <7 mcg yeast protein, and water for injection. The product does not contain a preservative or antibiotics.
  Gardasil-9 is supplied as a 0.5-mL single-dose vial or 0.5-mL single-dose prefilled Luer Lock syringe with tip cap. After thorough agitation, GARDASIL 9 is a white, cloudy liquid.
  Other Names: HPV Vaccine; 9-valent HPV vaccine (9vHPV)
Drug: Lidocaine injection — Lidocaine 1% will be injected intradermally and subcutaneously into the margin of the lymph node to be sampled to numb the area. To confer local anesthesia, 1-2% will be injected into the tissue surrounding the area where the bone marrow will be removed.
  Other Names: Lidocaine 1% Injectable Solution
Drug: Lorazepam — Lorazepam, an FDA-approved benzodiazepine, will be administered as an anxiolytic before the bone marrow aspirate procedure per the clinician who will perform the procedure. If needed, lorazepam will be administered sublingually per manufacturer dosing recommendations.

SUMMARY:
This study aims to answer the question: does 1-dose HPV vaccination generate the same immune responses compared to 2- or 3-dose HPV vaccination? This will be done by studying the immune response in blood, lymph nodes, and bone marrow.

Human papillomaviruses (HPV) cause cancers (cervical, anal, oropharyngeal, vulvar, vaginal, and penile), and the current HPV vaccine is highly effective at preventing disease by HPV types that cause 90% of cancer cases. While this vaccine generates high levels of antibodies that last for > 10 years, understanding of how this occurs is limited, and studying this immune response will help design new and better vaccines.

The study population consists of healthy adult (age 18-45) participants who have not previously received an HPV vaccine, do not have antibodies against certain types of HPV, do not have a history of HPV infection or disease (such as genital warts, abnormal pap test, or HPV DNA test), and do not have contraindications to study procedures. Populations of increased concern are not being enrolled.

DETAILED DESCRIPTION:
This study aims to determine whether a single-dose HPV vaccination produces the same immune response as a two- or three-dose HPV vaccination.

The 1-dose HPV vaccination was recently recommended by the World Health Organization (WHO) for people with healthy immune systems aged 9-20 years. To learn whether 1-dose HPV vaccination makes the same immune responses as 2- or 3-dose HPV vaccination in humans, there is a need to study the immune response to the HPV vaccine in the blood (where antibodies are), in the lymph nodes (where immune cells that make antibodies get activated), and in the bone marrow (where long-lived cells that produce antibodies are found). After informed consent, participants will have blood drawn for screening tests. If they are eligible, they will receive the FDA-approved HPV vaccine. The vaccine will be given in 1 or 2 doses, but participants will have the opportunity to receive the full vaccine series at the end of the study. Participants will have additional blood draws and undergo fine needle aspiration (FNA) of a lymph node in the axilla (armpit) at 3 different times. Later, they will have bone marrow aspiration procedures during which marrow is sampled from the hip bone through a needle. Researchers will use this knowledge to inform public health decisions about the broader use of 1-dose HPV vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-45 years old (inclusive), as the HPV vaccine is approved for this age range in adults
* BMI ≤ 32
* Able to understand and give informed consent (in American English).
* In good health based on physical examination, vital signs, medical history, and the investigator's clinical judgment.
* Available and willing to participate for the duration of this study
* Willing to undergo lymph node fine needle aspiration and bone marrow aspiration
* Willing to consent to the future use of remaining (residual) samples/specimens with IRB review
* Willing to defer completion of the recommended 9vHPV series

Exclusion Criteria:

* Ever received a dose of an HPV vaccine
* HPV 6, 11, 16, 18, 31, 33, 45, 52 or 58 seropositivity
* Any history of genital warts, an abnormal pap smear, or positive HPV DNA test
* Known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products
* Known allergy or history of anaphylaxis to yeast or products containing yeast.
* Any allergy to lidocaine.
* Pregnancy or breastfeeding.
* Participants who believe they cannot tolerate the lymph node fine needle aspirate or bone marrow aspirate procedures without general sedation
* Any history of lymphoma involving axillary nodes, any history of breast cancer, bilateral inflammatory process of upper arms in the past 2 weeks, prior breast or axillary biopsy and/or surgery that in the opinion of the investigator would affect the immune response results.
* Local infection, lymphadenitis, or rash in the targeted area.
* Received any vaccine from 14 days before the vaccine dose until 30 days after each vaccine dose* (*An individual initially excluded from study participation based on one or more of the time-limited exclusion criteria (fever, receipt of other vaccines) may be reconsidered for enrollment once the condition has resolved as long as the participant continues to meet all other entry criteria)
* Volunteers with fever (≥100.4 F or 38°C regardless of the route) within 3 days before vaccination*. (*An individual initially excluded from study participation based on one or more of the time-limited exclusion criteria (fever, receipt of other vaccines) may be reconsidered for enrollment once the condition has resolved as long as the participant continues to meet all other entry criteria)
* History of or presence of severe co-morbidities as determined by the investigator, including autoimmune disease, or clinically significant cardiac, pulmonary, gastrointestinal, hepatic, rheumatologic, renal disease, thrombocytopenia, and grade 4 hypertension** (**Grade 4 hypertension per CTCAE criteria is defined as life-threatening consequences (e.g., malignant hypertension, transient or permanent neurologic deficit, hypertensive)
* History of a bleeding disorder or currently taking anti-coagulant products*** (e.g. warfarin, direct thrombin inhibitors, heparin products, etc.), anti-platelet products, and/or NSAIDs including aspirin. (***including in the past week; however, an individual who is initially excluded from study participation based on one or more of the time-limited exclusion criteria may be reconsidered for enrollment once the condition has resolved as long as the participant continues to meet all other entry criteria)
* History of active malignancy other than squamous cell or basal cell skin cancer, unless there was a surgical excision considered to have achieved a cure.
* Current and/or expected immunosuppression due to cancer, receipt of chemotherapy, radiation therapy, and other immunosuppressive therapies (including anti-TNF therapy).
* Known or suspected congenital or acquired immunodeficiency, including functional or anatomic asplenia, or recent history or current use of immunosuppressive therapy****. (****Anti-cancer chemotherapy or radiation therapy within the preceding 3 years, or long-term (≥2 weeks within the previous 3 months) systemic corticosteroid therapy (e.g., prednisone at a dosage of ≥20 mg per day or on alternative days). Intranasal or topical prednisone (or equivalent) is allowed)
* Known chronic infections including, but not limited to, HIV, tuberculosis, hepatitis B or C.
* Is post-organ, bone marrow, and/or stem cell transplant, whether or not on chronic immunosuppressive therapy.
* Received blood products or immunoglobulin 3 months before study entry or planned use during this study.
* Had major surgery (per the investigator's judgment) within 4 weeks before study entry or planned major surgery during this study.
* Insulin-dependent diabetes***** mellitus type 1 or type 2 requiring therapy. (*****History of isolated gestational diabetes is not an exclusion criterion)
* Received experimental therapeutic agents within 12 months before the first vaccine dose or plans to receive any experimental therapeutic agents 12 months after the first vaccine dose that, at the investigator's discretion, would interfere with the safety or objectives of the study. COVID-19 vaccines that fall under FDA EUA will be treated as approved vaccines for this study.
* Is currently participating or plans to participate in another clinical study that would involve the receipt of an investigational product or undergo a procedure that, in the investigator's opinion would interfere with the safety or objectives of the study.
* Current diagnosed or self-reported alcohol abuse, drug abuse, or psychiatric conditions that in the opinion of the investigator would preclude compliance with the study.
* Social, occupational, or any other condition that in the investigator's discretion might interfere with compliance with the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Frequency of plasma cells specific for HPV16/18 virus like particles (VLPs) | 730 days after receiving the first vaccine dose
  Frequency of plasma cells specific for HPV16/18 virus-like particles (VLPs) per total IgG-secreting plasma cells in bone marrow in per-protocol participants of the 1- and 2-dose 9vHPV arms

SECONDARY OUTCOMES:
Frequency of memory B cells specific for HPV16/18 VLPs | Baseline (Day 0), Day 30, Day 180, Day 210, Day 365, and Day 730 post-intervention
  Frequency of memory B cells specific for HPV16/18 VLPs per total memory B cells in PBMC in per protocol participants of the 1- and 2-dose 9vHPV arms.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Scherer, PhD, Principal Investigator — Emory University
Locations (1):
- Hope Clinic of the Emory Vaccine Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share de-identified demographic, ELISPOT, pseudovirus neutralization, ELISA, flow cytometry, sc-RNA-seq, paired immunoglobulin repertoire sequencing, monoclonal antibody neutralization, and the monoclonal antibody heavy and light chain sequence data utilized in our publications. Data will be made publicly available in relevant repositories and easy to find in their publications.
Supporting Information: Study Protocol, ICF
Time Frame: Available immediately following publication. No end date.
Access Criteria: De-identified data will be published in an open-access journal with no access restrictions; De-identified RNA-seq data will be deposited at public repositories with no access restrictions.